CLINICAL TRIAL: NCT03198299
Title: Therapeutic Effects of Physical Function and Balance of Arch Support Insoles on Children
Brief Title: Therapeutic Effects of Arch Support Insoles on Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, primary investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SKH-8302-105-DR-24
Record Dates: First submitted 2017-06-13; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Normal Development
Keywords: therapeutic effects; insoles; children

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group: MEI BIN insoles (Active Comparator): Study group: participants in the study group were prescribed with customized insoles (MEI BIN insoles) to keep the subtalar joint in neutral position, for 12 weeks.
  Interventions: Device: MEI BIN insoles
- control group: without MEI BIN insoles (No Intervention): Control group: participants in the control group were not prescribed with customized insoles (MEI BIN insoles) to keep the subtalar joint in neutral position, for 12 weeks.

INTERVENTIONS:
Device: MEI BIN insoles — wearing insoles for 12 weeks
  Arms: study group: MEI BIN insoles

SUMMARY:
Using double blind, randomized controlled design to study the short-term therapeutic effects of customized arch support insoles on children

DETAILED DESCRIPTION:
A total of 45 children were enrolled. The children were randomized into two groups, including the study group (insoles group) and the control group (without insoles group).

All participants in the insoles group were evaluated at baseline, that was before the customized arch-support insoles were prescribed. All the evaluations, including functional performance, physical function, and quality of life, were re-evaluated up to 12 weeks after the insoles wearing in the study group (insoles group).

The control group were evaluated at baseline and up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* children with age 3 to 10 can walk independently for 15 meters can follow up for 12 weeks

Exclusion Criteria:

* age less than 3 years or older than 10 years children with developmental delays children with pathological flat feet

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
change of baseline of level walking time to 12 weeks | baseline and up to 12 weeks
  time of level walking
change of baseline of stairs climbing time to 12 weeks | baseline and up to 12 weeks
  time of stairs climbing
change of baseline of up and go time to 12 weeks | baseline and up to 12 weeks
  time of up and go
change of baseline of chair raising time to 12 weeks | baseline and up to 12 week
  time of chair raising

SECONDARY OUTCOMES:
change of baseline balance (scores) to 12 weeks | baseline and up to 12 weeks
  Berg balance test
change of baseline functional performance(scores) to 12 weeks | baseline and up to 12 weeks
  Pediatric Outcome Data Collection instrument
change of baseline quality of life (scores) to 12 weeks | baseline and up to 12 weeks
  Child Health Questionnaire-Parent form

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No